CLINICAL TRIAL: NCT04215406
Title: The Effects of Maternal Exposure to Air Pollution During Pregnancy on Adverse Pregnancy Outcomes Mediated by Inflammatory Cytokine and Hormone
Brief Title: The Mechanism of Adverse Pregnancy Outcomes Influenced by Maternal Air Pollution Exposure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2019-023
Record Dates: First submitted 2019-12-25; First posted 2020-01-02 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2021-08

CONDITIONS: Adverse Pregnancy Outcomes
Keywords: pregnancy; air pollution; inflammatory cytokine; hormone; effect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The venous blood from pregnant women is acquired in different time point for measurement of serum concentration of inflammatory cytokine and hormone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The level of maternal air pollution exposure during pregnancy: The groups will be decided according to the level of maternal exposure to air pollution during pregnancy. Participants will be divided into experimental group (high level of maternal air pollution exposure) and control group (low level of maternal air pollution exposure) or other groups according to research and actual demand.
  Interventions: Other: The level of air pollution

INTERVENTIONS:
Other: The level of air pollution — The intervention measure is the level of air pollution, it is a non-human interventional measure based on the weighted average of various air pollutants monitored by air pollution monitoring stations during different period of pregnancy.

SUMMARY:
This research evaluates the effects of maternal exposure to air pollution during pregnancy on adverse pregnancy outcomes, the general demographic information, the level of maternal exposure to air pollution, pregnancy-related information, the occurrence of adverse pregnancy outcomes, and serum indicators of pregnant women during pregnancy are collected. Finally, the research explores that whether the inflammatory cytokine and hormone can mediate the occurrence of adverse pregnancy outcomes under the maternal exposure to air pollution during pregnancy.

DETAILED DESCRIPTION:
Pregnancy is the most important period in the life process. China have a high occurrence of adverse pregnancy outcomes and the situation of air pollution is not optimistic. With the introduction of perspective in environment and health, the impact of air pollution on health has received extensive attention. A large number of studies have confirmed that maternal exposure to air pollution during pregnancy such as particulate matter (PM), nitrogen dioxide (NO2), sulfur dioxide (SO2), ozone (O3), carbon monoxide (CO) can increase the risk of miscarriage, gestational diabetes mellitus(GDM), hypertensive disorder complicating pregnancy, preterm birth and low birth weight(LBW). Maternal exposure to air pollution was also closely related to birth defects, newborn congenital hypothyroidism, and affect neurodevelopment in offspring. In other respects, studies shown that air pollution can change maternal steroid hormone levels (human chorionic gonadotropin (hCG), luteinizing hormone (LH), follicle-stimulating hormone (FSH), estradiol(E2) and progesterone(P)), which play an important role in maintaining pregnancy and the developing of adverse pregnancy outcomes. Interleukin (IL) is an important inflammatory mediator cytokine, IL-8, IL-6 and IL-2 are closely related to the reproductive process of mammals and may regulate the occurrence of adverse pregnancy outcomes and influenced by air pollution, but limited studies focused on them in regulating the occurrence of adverse pregnancy outcomes under exposure to air pollution. So, a prospective cohort study is conducted to explore the new mechanism of adverse pregnancy outcomes affected by air pollution.

Research content: This research is a prospective cohort study from January 2020 to December 2022, 288 pregnant women will be recruited from the First Affiliated Hospital of Xi'an Jiaotong University. A health management birth cohort will be established. The subjects will be enrolled within 6 weeks of gestation, and be followed up about 9 months: ①To construct a spatial and temporal series about adverse pregnancy outcomes influenced by maternal exposure to air pollution during pregnancy; ②To explore the effects of maternal exposure to air pollution on hormone and inflammatory cytokine during pregnancy, and the relationship between maternal level of hormone, inflammation cytokine and adverse pregnancy outcomes; ③To determine if maternal hormone and inflammatory cytokine mediate the occurrence of adverse pregnancy outcomes during pregnancy under maternal exposure to air pollution as intermediate regulatory product.

Research meaning：①To explore the mechanism of adverse pregnancy outcomes affected by air pollution during pregnancy, provide an epidemic evidence for interposing the occurrence of adverse pregnancy outcomes by regulating maternal hormone and inflammatory cytokine; ②To define the critical period of the developing of adverse pregnancy outcomes in spatial and temporal series, and to calculate the cutoff value of air pollution on adverse pregnancy outcomes, propose short-term control target of air pollution related to maternal and child health, construct the first-level prevention strategy for adverse pregnancy outcomes.

Research steps: ① Complete the recruiting of subjects, which meet the inclusion and exclusion criteria sign an informed consent before the carrying out of research; ② Follow up: Three questionnaires will be conducted at the end of each trimester to acquire the information including sociodemographic characteristics, menstrual history and childbearing history, residence during pregnancy, lifestyle and diet habits, the information of illness and medication, history of past illness, etc. Then the maternal exposure level of air pollutants in every trimester will be calculated, based on air pollution detection station, from Shaanxi Meteorological and Environment Bureau according to residence information of participants; ③ Serum indicators: fasting venous blood samples will be taken at different time points to detect serum level of maternal hormone and inflammatory cytokine, all the venous blood samples will be taken and tested in the laboratory of First Affiliated Hospital of Xi'an Jiaotong University. 4 mL of fasting venous blood sample are needed, and the blood sample will be put in dry test tubes, centrifuged within 1 hour, and the separated serum was stored at -20 ° C, chemiluminescence and ELASA will be adapted to detect the samples respectively. ④ Monitoring of adverse pregnancy outcomes: closely monitor the occurrence of adverse pregnancy outcomes during pregnancy. During the whole study period, the subjects could withdraw the cohort at any time.

Abortion: The abortion includes early spontaneous abortion (occur within 12 weeks of gestation), late spontaneous abortion (occur from 12 weeks to 28 weeks of gestation) and missed abortion included(embryo die in the uterine cavity and fail to excrete themselves at time); Maternal adverse pregnancy outcomes: hypertension disorders of pregnancy (gestational hypertension, preeclampsia, eclampsia, chronic hypertension), GDM (referring to diabetes occur in pregnancy and the glucose metabolism is normal before pregnancy). Adverse outcomes for fetus or newborn: including preterm birth (delivery form 28 weeks to 37 weeks of gestation); low birth weight (newborn weight measured within 72 hours after birth is less than 2500 grams); birth defects (fetal structural, functional or metabolic abnormalities, also known as congenital malformations).

Statistical method: ①Univariate analysis: The maternal exposure levels of air pollution during pregnancy will be treated as independent variables, pregnancy outcomes will be treated as dependent variables, univariate logistic regression will be used to analyze the relationship between them; Then, maternal exposure levels will be treated as independent variables, maternal hormone and inflammatory cytokine as the dependent variable, the univariate logistic regression analysis will be used to analyze the relationship between them; Finally, the level of hormone and inflammatory cytokine will be treated as independent variables, pregnancy outcomes as dependent variables, and analyze the relationship between them; ②Multivariate analysis: adverse pregnancy outcomes will be taken as dependent variables, maternal exposure levels, sociodemographic characteristics, nutritional status, dietary status, and other factors are included as independent variables, the multivariate logistic regression analysis will be used to data analysis. In the multivariate regression the odds ration value and 95% confidence intervention of air pollution to affect adverse pregnancy outcomes will be calculated adjusted for sociodemographic characteristics, nutrition, dietary conditions and other factors; ③Analysis of intermediary factor: mediate effect analysis will be used to analyze whether the maternal hormone and inflammatory cytokine mediate the occurrence of adverse pregnancy outcomes as intermediate regulatory products under maternal air pollution exposure; ④ Spatial and temporal series analysis will be adapted to define the critical period of the developing of adverse pregnancy outcomes under maternal exposure to air pollution, and calculate the cut-off value of air pollution about the adverse pregnancy outcomes.

Research planning: ①Complete research design, follow-up questionnaires, and pre-experiments before 2020; ②Complete enrollment of subjects, follow-up of the study subjects, detecting of serum indicators, monitor the occurrence of adverse pregnancy outcomes before January 2021; ③Complete data export and analysis about basic information and data analysis; ④Clarify the relationship between maternal air pollution exposure during pregnancy and adverse pregnancy outcomes, explore the potential mechanism in the occurrence of adverse pregnancy outcomes influenced by air pollution.

ELIGIBILITY:
Inclusion Criteria:

* The Pregnant women within 6 weeks of gestation from the First Affiliated Hospital of Xi'an Jiaotong University;
* This pregnancy is natural conception, the last menstrual period is definite and the menstrual cycle is basically regular;
* The pregnant examinations are performed in our hospital;
* The pregnant women volunteer to participate in this study and sign the informed consent.

Exclusion Criteria:

* The couples have chromosomal abnormalities or hereditary diseases;
* The pregnant women have trophoblastic diseases such as hydatidiform mole;
* The pregnant women with genital malformations, such as mediastinal uterus, single-horned uterus, double uterus, etc;
* The pregnant women are definitively diagnosed with uterine fibroids, ovarian cysts, polycystic ovary syndrome, gynecological inflammation and other gynecological diseases;
* The pregnant women are definitively diagnosed with hypertensive, diabetes and other chronic disease before pregnancy;
* The pregnant women are definitively diagnosed with autoimmune diseases such as systemic lupus erythematosus, multiple arteriolar inflammation, rheumatoid arthritis, etc;
* The participants have other serious diseases.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study participants are healthy pregnant women within 6 weeks of pregnancy from the First Affiliated Hospital of Xi'an Jiaotong University, who meet the inclusion and exclusion criteria, and sign the informed consent before the implementation of this research. All the participants will be followed up about 9 months and measured the serum concentration of inflammatory cytokine and hormone.
Sampling Method: Probability Sample
Enrollment: 288 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The occurrence of adverse pregnancy outcomes or delivery | ①For abortion, up to 24 weeks. ②For participants without abortion will be assessed when hypertension disorders of pregnancy and GDM occur, then assessment of preterm birth, LBW and birth defects will be conducted when delivery, up to about 9 months
  Adverse pregnancy outcomes including abortion, gestational diabetes mellitus (GDM), hypertensive disorder complicating pregnancy, preterm birth, birth defects and low birth weight(LBW).

CONTACTS AND LOCATIONS:
Overall Officials: Wenfang Yang, PHD, Study Director — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No